CLINICAL TRIAL: NCT07165301
Title: Prospective Cohort Study of Functional Dyspepsia/Postprandial Distress Syndrome Patients Treated With Itopride
Brief Title: Postprandial Distress Itopride Cohort Trial
Acronym: PASSPORT
Status: Not yet recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S70891
Record Dates: First submitted 2025-08-20; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Postprandial Distress Syndrome; Functional Dyspepsia; Epigastric Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Functional dyspepsia patients

SUMMARY:
Functional Dyspepsia (FD) is a common gastrointestinal disorder affecting about 7.2% of the population, characterized by gastroduodenal symptoms without an identifiable organic cause. It is divided into two subtypes based on the Rome IV criteria: (i) Postprandial Distress Syndrome (PDS): Meal-related symptoms like postprandial fullness and early satiation.; (ii) Epigastric Pain Syndrome (EPS): Meal-unrelated symptoms like epigastric pain or burning.

Treatment options are limited, but prokinetics are commonly used, targeting suspected motility issues. A meta-analysis showed prokinetics reduce symptoms. Itopride, a D2 antagonist and acetylcholinesterase inhibitor, has shown potential efficacy, especially in Asian populations.

As Itopride became available in Belgium since 2023, there is a lack of real-life outcome data in Western patients with functional dyspepsia/postprandial distress syndrome who receive treatment in standard clinical practice. Hence, the aim of this pragmatic observational study is to follow up a cohort of functional dyspepsia/postprandial distress syndrome patients in whom itopride treatment is started as part of routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with functional dyspepsia as per physician clinical criteria
* Patient must sign an informed consent document before the initiation of any study-related procedures indicating that he or she understands the purpose and procedures required for the study and is willing to participate in the study.
* Patient must speak Dutch or French

Exclusion Criteria:

* Patient with other clinical diagnosis than functional dyspepsia that can explain their gastrointestinal symptoms.
* Patient has any of the following surgical history:

  * Any abdominal surgery within the 3 months prior to screening;
  * Subject has a history of major gastric, hepatic, pancreatic, or intestinal surgery (appendectomy, hemorrhoidectomy, cholecystectomy, or polypectomy more than 3 months earlier are allowed).
* Patient has an unstable cardiac, pulmonary, renal, hepatic, metabolic, or hematologic condition.
* Patient has a history of active malignancy within 3 years before screening (except squamous and basal cell carcinomas and cervical carcinoma in situ).
* Patient has received an investigational drug or used an investigational medical device within 30 days prior to randomization, or is currently enrolled in an investigational study.
* In case of psychotropic drug use: patient NOT on stable doses of antidepressants (i.e., for the 3 months prior to pre-screening) will not be allowed to participate in the study. Habitual use of benzodiazepines is permitted.
* Patient is pregnant or breastfeeding.
* Patient has any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are recruited in Belgium at gastroenterology outpatient clinics when their treating gastroenterologist decides to initiate itopride as part of standard clinical care for functional dyspepsia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
PAGI-SYM improvement | 8 weeks
  The primary endpoint for this study is symptom improvement at week 8. For this, the symptomatic improvement as assessed by the Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) compared to baseline will be evaluated for each symptomatic domain (heartburn/regurgitation, fullness/early satiety, nausea/vomiting, bloating, upper abdominal pain, lower abdominal pain) where a MCID has been previously been established.

SECONDARY OUTCOMES:
Symptom Improvement | From baseline to +16 weeks (end of trial)
  Symptom evolution will be assessed using the PAGI-SYM questionnaire. The PAGI-SYM will be administered at baseline, week 8, and week 16 to evaluate changes in individual gastrointestinal symptoms over time. Previously established minimal clinically important differences (MCIDs) will be used to aid in the interpretation of changes.
Perceived Treatment Effectiveness | From baseline to +16 weeks (end of trial)
  Perceived treatment effectiveness will be assessed using the Overall Treatment Evaluation (OTE) questionnaire. The OTE will be assessed at visit 1 and visit 2 to capture the patient's subjective sense treatment effectiveness. Together with the PAGI-SYM questionnaire, these instruments will provide both objective and patient-perceived measures of symptom change during the study period.
Health-economic evaluation: WPAI | -6 months to +16 weeks (end of trial)
  Health-economic outcomes will be assessed using the Work Productivity and Activity Impairment (WPAI) questionnaire. This instrument will be used to evaluate changes in work productivity related to gastric symptoms. Together with the EuroQol 5 Dimension 5 Level (EQ-5D-5L) and Health Resource Utilization (HRU) questionnaires, these data will be used to assess the economic impact of the intervention.
Health-economic evaluation and quality of life: EQ-5D-5L | -6 months to +16 weeks (end of trial)
  Health-economic outcomes and quality of life will be assessed using the EQ-5D-5L questionnaire. This instruments will be used to evaluate changes in health-related quality of life related to gastric symptoms. Quality-adjusted life years (QALYs) will be calculated based on EQ-5D-5L responses to support cost-utility analysis.
Health-economic evaluation: HRU | -6 months to +16 weeks (end of trial)
  Health-economic outcomes will be assessed using the HRU questionnaire. This instrument will be used to evaluate changes in healthcare resource utilization related to gastric symptoms.Health resource use will be collected retrospectively for the 6 months prior to baseline and prospectively throughout the study to estimate direct medical costs.
Quality of life evaluation | From baseline to +16 weeks (end of trial)
  Quality of life will be assessed using the Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QOL) questionnaire at baseline, week 8, and week 16. This instrument will be used to evaluate the specific impact of gastrointestinal symptoms on daily functioning and well-being.
Treatment compliance | From +8 weeks to +16 weeks (end of trial)
  Treatment adherence will be assessed through self-report, and expressed as the proportion of prescribed doses taken during the study period. Compliance will be analyzed descriptively and explored as a potential factor influencing treatment outcomes.
Baseline characteristics | From baseline to +16 weeks (end of trial)
  Baseline characteristics include medical history and demographic parameters (age, sex, weight, length, BMI). Baseline economic impact will be assessed by the Health resource utilisation (HRU) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided